CLINICAL TRIAL: NCT03973177
Title: Phenol Neurolysis of Genicular Nerves for Chronic Knee Pain Following Total Knee Arthroplasty: a Pilot Prospective, Randomized, Crossover Trial
Brief Title: Phenol Neurolysis of Genicular Nerves for Chronic Knee Pain
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Covid restrictions on recruitment
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, David Walega, Principal Investigator, Northwestern University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: STU00209591
Record Dates: First submitted 2019-05-28; First posted 2019-06-04 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2022-04

CONDITIONS: Pain, Chronic
Keywords: Total knee arthroplasty; Chronic Pain
MeSH Terms: conditions — Chronic Pain | interventions — Phenol; Methylprednisolone; Methylprednisolone Acetate

STUDY DESIGN:
Intervention Model Description: A Pilot Prospective, Randomized, Crossover Trial. (Block randomization scheme with 2:1 allocation (phenol neurolysis : perineural steroid injection) The crossover will occur in subjects who received the steroid injection who did not achieve adequate pain relief at 3 months.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment Group: Phenol injection (Experimental): 6% aqueous phenol 2.5 mL will be mixed with 0.5 mL iopamidol 300 and will be injected at each target sites
  Interventions: Drug: Phenol Injection
- Control Group: Methylprednisolone injection (Other): Methylprednisolone acetate 10 mg with 2 mL preservative free saline and 0.5 mL iopamidol 300 will be injected at each of the target site
  Interventions: Drug: Methylprednisolone Injection

INTERVENTIONS:
Drug: Phenol Injection — 6% aqueous phenol 2.5 mL will be mixed with 0.5 mL iopamidol 300 and will be injected at each target site with live, pulsed fluoroscopy (5-8 seconds at each location) to observe the contrast dye-tagged phenol covering the lateral margin of the femur or tibia respectively on AP and lateral views. The needles will then be removed and band-aids placed.
  Other Names: Phenol
  Arms: Treatment Group: Phenol injection
Drug: Methylprednisolone Injection — Methylprednisolone acetate 10 mg with 2 mL preservative saline and 0.5 mL iopamidol 300 will be injected at each of the 3 target sites with live, pulsed fluoroscopy (5-8 seconds at each location) to observe the contrast dye-tagged steroid mixture covering the lateral margin of the femur or tibia respectively on AP and lateral views; the needles will be removed and band-aids placed.
  Other Names: Methylprednisolone acetate
  Arms: Control Group: Methylprednisolone injection

SUMMARY:
Chronic knee pain from osteoarthritis (OA) is commonly treated with total knee arthroplasty (TKA) when conservative therapies fail to provide pain relief. More than 600,000 TKAs are performed in the U.S. annually, a number that continues to increase. A logistic-regression model suggests that the incidence rate of TKA will increase by 143% in the United States by 2050 compared to 2012. Although TKA is successful in reducing knee pain and joint stiffness in most cases, it can be associated with a 7-35% incidence of persistent refractory post-surgical knee pain.

Aim:

To determine whether chemical neurolysis of the genicular nerves with 6% aqueous phenol is non-inferior in reducing knee pain as compared to corticosteroid injection of the genicular nerves, in patients with refractory chronic knee pain for more than 6 months after total knee replacement.

Hypothesis:

Chemical neurolysis of genicular nerves with phenol will provide equal or superior pain relief than corticosteroid genicular nerve injections at 3 months, as measured by the Oxford Knee Score.

ELIGIBILITY:
Inclusion Criteria:

* Ages 40-95 years
* Patients with knee pain, on average > 4 (NRS) persisting more than 6 months after TKA
* Willingness to undergo image guided diagnostic nerve block and the study intervention

Exclusion Criteria:

* Pain score (NRS) < 4 at time of study enrollment
* Conditions that preclude the diagnostic block or the study intervention (e.g., irreversible coagulopathy or bleeding disorder, allergic reaction/contraindication to local anesthetic, contrast dye, steroids, and/or phenol, pregnancy, severe or uncontrolled medical illness).
* Evidence of indolent infection of the knee prosthesis (elevated C-reactive protein assessed when clinically indicated)
* Inability to write, speak, or read in English
* Pregnancy

Ages: 40 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-05-24 (Actual); Primary Completion 2022-07 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Oxford Knee Score | 3 months
  Oxford Knee Score is a tool which measures 6 post operative items (pain,flexion contracture, extension lag, total range of flexion, alignment of varus and valgus,stability (antero-posterior and mediolateral). The scoring is: below 60 is poor, scoring 60-69 fair, scoring 70-79 good, 80-100 excellent.

SECONDARY OUTCOMES:
Numeric Rating Scale Score | 3months
  The proportion of subjects who have > 50% reduction in pain based on the Numeric Rating Scale at 3 months. The NRS is a scale of 0 (no pain) to 10 (worst pain imaginable)
Numeric Rating Scale Score | 6 months
  The proportion of subjects who have > 50% reduction in pain based on the Numeric Rating Scale at 6 months. The NRS is a scale of 0 (no pain) to 10 (worst pain imaginable)
Patients Global Impression of Change | 3 Months
  Patients Global Impression of Change (GPIC) is a scale of 0 (much better) to 10 (much worse)
Patients Global Impression of Change | 6 Months
  Patients Global Impression of Change (GPIC) is a scale of 0 (much better) to 10 (much worse)
Opioid analgesic use at 3 months | 3 months
  Opioid analgesic daily use by self reporting .
Opioid analgesic use at 6 months | 6 months
  Opioid analgesic daily use by self reporting.
Non-opioid analgesic use at 3 months | 3 Months
  Non opioid analgesic daily use by self reporting.
Non-opioid analgesic use at 6 months | 6 Months
  Non opioid analgesic daily use by self reporting.
PROMIS Pain Intensity Short Form 3a | Baseline
  3 question pain survey. 5 responses (had no pain),(mild), (moderate), (severe) and (very severe)
PROMIS Pain Intensity Short Form 3a | 3 Months
  3 question pain survey. 5 responses (had no pain),(mild), (moderate), (severe) and (very severe)
PROMIS Pain Intensity Short Form 3a | 6 Months
  3 question pain survey. 5 responses (had no pain),(mild), (moderate), (severe) and (very severe)
PROMIS Sleep Disturbance Short Form 4a | Baseline
  4 question sleep survey. First section is quality of sleep rated on a 5 response (very poor)- (very good) scale.Section rating quality of sleep based on 5 response choices (not at all) to (very much)
PROMIS Sleep Disturbance Short Form 4a | 3 Months
  4 question sleep survey. First section is quality of sleep rated on a 5 response (very poor)- (very good) scale.Section rating quality of sleep based on 5 response choices (not at all) to (very much)
PROMIS Sleep Disturbance Short Form 4a | 6 Months
  4 question sleep survey. First section is quality of sleep rated on a 5 response (very poor)- (very good) scale.Section rating quality of sleep based on 5 response choices (not at all) to (very much)
PROMIS Pain Interference Short Form 6b | Baseline
  6 question pain survey. First section is interference of pain rated on a 5 response (not at all)- (very much) scale. Section is one socialization question with 5 response choices (never)- (always)
PROMIS Pain Interference Short Form 6b | 3 Months
  6 question pain survey. First section is interference of pain rated on a 5 response (not at all)- (very much) scale. Section is one socialization question with 5 response choices (never)- (always)
PROMIS Pain Interference Short Form 6b | 6 Months
  6 question pain survey. First section is interference of pain rated on a 5 response (not at all)- (very much) scale. Section is one socialization question with 5 response choices (never)- (always)
Oxford Knee Score | Baseline
  12 question survey with 5 choice responses based on severity of pain while accomplishing activities of daily living.
Oxford Knee Score | 6 Months
  12 question survey with 5 choice responses based on severity of pain while accomplishing activities of daily living.
Hospital Anxiety and Depression Scale | Baseline
  Hospital Anxiety and Depression Scale (HADS) is a 14 question survey (7 anxiety and 7 depression) questions answered on a 0 (low) - 3 (high) scale.Total score of 0-7 is normal, 8-10 is baseline abnormal and a score between 11-21 is abnormal.
Hospital Anxiety and Depression Scale | 3 Month
  Hospital Anxiety and Depression Scale (HADS) is a 14 question survey (7 anxiety and 7 depression) questions answered on a 0 (low) - 3 (high) scale.Total score of 0-7 is normal, 8-10 is baseline abnormal and a score between 11-21 is abnormal.
Hospital Anxiety and Depression Scale | 6 Month
  Hospital Anxiety and Depression Scale (HADS) is a 14 question survey (7 anxiety and 7 depression) questions answered on a 0 (low) - 3 (high) scale. Total score of 0-7 is normal, 8-10 is baseline abnormal and a score between 11-21 is abnormal.

CONTACTS AND LOCATIONS:
Overall Officials: David Walega, MD, Principal Investigator — Northwestern University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nguyen US, Zhang Y, Zhu Y, Niu J, Zhang B, Felson DT. Increasing prevalence of knee pain and symptomatic knee osteoarthritis: survey and cohort data. Ann Intern Med. 2011 Dec 6;155(11):725-32. doi: 10.7326/0003-4819-155-11-201112060-00004. PMID 22147711
- [Background] Buvanendran A, Fiala J, Patel KA, Golden AD, Moric M, Kroin JS. The Incidence and Severity of Postoperative Pain following Inpatient Surgery. Pain Med. 2015 Dec;16(12):2277-83. doi: 10.1111/pme.12751. Epub 2015 Apr 27. PMID 25917518
- [Background] Lewis GN, Rice DA, McNair PJ, Kluger M. Predictors of persistent pain after total knee arthroplasty: a systematic review and meta-analysis. Br J Anaesth. 2015 Apr;114(4):551-61. doi: 10.1093/bja/aeu441. Epub 2014 Dec 26. PMID 25542191
- [Background] Drosos GI, Triantafilidou T, Ververidis A, Agelopoulou C, Vogiatzaki T, Kazakos K. Persistent post-surgical pain and neuropathic pain after total knee replacement. World J Orthop. 2015 Aug 18;6(7):528-36. doi: 10.5312/wjo.v6.i7.528. eCollection 2015 Aug 18. PMID 26301182
- [Background] Puolakka PA, Rorarius MG, Roviola M, Puolakka TJ, Nordhausen K, Lindgren L. Persistent pain following knee arthroplasty. Eur J Anaesthesiol. 2010 May;27(5):455-60. doi: 10.1097/EJA.0b013e328335b31c. PMID 20299989
- [Background] Fischer HB, Simanski CJ, Sharp C, Bonnet F, Camu F, Neugebauer EA, Rawal N, Joshi GP, Schug SA, Kehlet H; PROSPECT Working Group. A procedure-specific systematic review and consensus recommendations for postoperative analgesia following total knee arthroplasty. Anaesthesia. 2008 Oct;63(10):1105-23. doi: 10.1111/j.1365-2044.2008.05565.x. Epub 2008 Jul 10. PMID 18627367
- [Background] Inacio MCS, Paxton EW, Graves SE, Namba RS, Nemes S. Projected increase in total knee arthroplasty in the United States - an alternative projection model. Osteoarthritis Cartilage. 2017 Nov;25(11):1797-1803. doi: 10.1016/j.joca.2017.07.022. Epub 2017 Aug 8. PMID 28801208
- [Background] Sylvester LN, Goree JH. Genicular Radiofrequency Ablation for Treatment of Post Total Knee Arthroplasty Posterior Thigh Pain: A Case Report. A A Case Rep. 2017 Nov 15;9(10):292-293. doi: 10.1213/XAA.0000000000000596. PMID 28697032
- [Background] Qudsi-Sinclair S, Borras-Rubio E, Abellan-Guillen JF, Padilla Del Rey ML, Ruiz-Merino G. A Comparison of Genicular Nerve Treatment Using Either Radiofrequency or Analgesic Block with Corticosteroid for Pain after a Total Knee Arthroplasty: A Double-Blind, Randomized Clinical Study. Pain Pract. 2017 Jun;17(5):578-588. doi: 10.1111/papr.12481. Epub 2016 Sep 19. PMID 27641918
- [Background] Protzman NM, Gyi J, Malhotra AD, Kooch JE. Examining the feasibility of radiofrequency treatment for chronic knee pain after total knee arthroplasty. PM R. 2014 Apr;6(4):373-6. doi: 10.1016/j.pmrj.2013.10.003. Epub 2013 Dec 27. PMID 24373908
- [Background] Walega DR, McCormick ZL. Chemical Neurolysis of the Genicular Nerves for Chronic Knee Pain: Reviving an Old Dog and an Old Trick. Pain Med. 2018 Sep 1;19(9):1882-1884. doi: 10.1093/pm/pny023. No abstract available. PMID 29514315
- [Background] Koyyalagunta D, Engle MP, Yu J, Feng L, Novy DM. The Effectiveness of Alcohol Versus Phenol Based Splanchnic Nerve Neurolysis for the Treatment of Intra-Abdominal Cancer Pain. Pain Physician. 2016 May;19(4):281-92. PMID 27228515
- [Background] Wang PJ, Shang MY, Qian Z, Shao CW, Wang JH, Zhao XH. CT-guided percutaneous neurolytic celiac plexus block technique. Abdom Imaging. 2006 Nov-Dec;31(6):710-8. doi: 10.1007/s00261-006-9153-5. PMID 17151902
- [Background] Kirazli Y, On AY, Kismali B, Aksit R. Comparison of phenol block and botulinus toxin type A in the treatment of spastic foot after stroke: a randomized, double-blind trial. Am J Phys Med Rehabil. 1998 Nov-Dec;77(6):510-5. doi: 10.1097/00002060-199811000-00012. PMID 9862538
- [Background] Ahmed A, Arora D, Kochhar AK. Ultrasound-guided alcohol neurolysis of lateral femoral cutaneous nerve for intractable meralgia paresthetica: a case series. Br J Pain. 2016 Nov;10(4):232-237. doi: 10.1177/2049463716668811. Epub 2016 Sep 16. PMID 27867513